CLINICAL TRIAL: NCT05678049
Title: Evaluation and Characterisation of Microplastics and Nanoplastics in Joint Synovial Liquid
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Ciubean Alina Deniza, Director, Iuliu Hatieganu University of Medicine and Pharmacy
Other Study IDs: UMFCluj
Record Dates: First submitted 2022-12-15; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Osteoarthritis, Knee; Knee Arthritis; Gout Arthritis; Microcrystal Disease
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis, Gouty; Elephantiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Synovial fluid analysis — For patients with knee under tension at the joint level, the symptomatology often requires evacuation by puncture under ultrasound guidance. The intervention will be performed only for patients for whom this therapeutic indication exists anyway by their physicians.
  After making the evacuation we will want to use this liquid for Microscopic and Spectrophotometric evaluation

SUMMARY:
The research study aims to evaluate the synovial fluid to highlight the presence of possible micropolymers (micro/nanoplastics) in order to better understand the pathophysiology of joint degenerative processes. For patients with liquid under tension at the joint level, the symptomatology often requires evacuation by puncture under ultrasound guidance. The intervention will be performed only for patients for whom this therapeutic indication exists anyway by their physician.

The investigators want to use this liquid for Microscopic and Spectrophotometric evaluation.

ELIGIBILITY:
Inclusion Criteria:

* arthritis of the knee with liquid aspiration recommendation
* age >18 years

Exclusion Criteria:

--refusal of the patient to participate

-age<18 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients on a Rehab Department with arthritis of the knee that require evacuation of the knee joint
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
microplastics | immediately after liquid extraction
  evaluation with spectrophotometry and optic microscopy
nanoplastics | immediately after liquid extraction
  evaluation with spectrophotometry and optic microscopy